CLINICAL TRIAL: NCT00042458
Title: A Randomized, Triple-Blind, Placebo-Controlled, Multicenter Study to Investigate the Safety of Pramlintide Treatment Employing Pramlintide Dose-Titration Followed by Insulin Dose Optimization in Subjects With Type 1 Diabetes Mellitus Who Have Not Achieved Glycemic Targets With Intensive Insulin Therapy
Brief Title: Evaluation of Dose-titration of Pramlintide During Initiation of Therapy in Patients Trying to Improve Glucose Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 137-150
Record Dates: First submitted 2002-07-30; First posted 2002-08-01 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — pramlintide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo injection will be supplied in the same 5-mL multidose glass vials with a rubber stopper.Ingredients: D-Mannitol 43.0 mg/mL Metacresol 2.25 mg/mL Glacial acetic acid 1.53 mg/mL Sodium acetate trihydrate 0.61 mg/mL pH 4.0 Water for injection qs to 5.0 mL
  Interventions: Drug: Placebo
- Pramlintide Acetate (AC137) (Active Comparator): Pramlintide acetate (AC137) injection is a clear, colorless, sterile solution for SC injection. It consists of pramlintide in sodium acetate buffer, pH 4.0, containing 43 mg/mL mannitol as an iso-osmolality modifier and 2.25 mg/mL metacresol as a preservative. The strength of pramlintide injection is 0.6 mg/mL
  Interventions: Drug: Pramlintide acetate

INTERVENTIONS:
Drug: Pramlintide acetate — Pramlintide injection will be supplied in 5-mL multidose glass vials with rubber stoppers.
  Arms: Pramlintide Acetate (AC137)
Drug: Placebo — The placebo injection will be supplied in the same 5-mL multidose glass vials with a rubber stopper.
  Arms: Placebo

SUMMARY:
This is a randomized, triple-blind, placebo-controlled, multicenter study to investigate the safety of pramlintide treatment using pramlintide dose-titration coupled with insulin adjustments in subjects with type 1 diabetes who are actively trying to improve their glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c value between 7.5-9%
* Using multiple daily insulin injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2002-04; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
- To investigate the safety of pramlintide treatment employing dose titration upon initiation of pramlintide followed by insulin dose optimization in subjects with type 1 diabetes. | 29 Weeks

SECONDARY OUTCOMES:
- To examine the change in HbA1c, postprandial glucose concentration, and body weight over the course of the study. | 29 Weeks
- To examine the pattern of daily insulin use over the course of the study. | 29 Weeks

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Ana Ventures LLC, Mesa, Arizona
  - Phoenix Endocrinology Clinic, Ltd., Phoenix, Arizona
  - East Bay Clinical Trial Center, Concord, California
  - Valley Research, Fresno, California
  - UCSD Diabetes Research Center, San Diego, California
  - Diabetes Research Institute, San Mateo, California
  - Sansum Medical Research Institute, Santa Barbara, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center for Childhood Diabetes, Denver, Colorado
  - MedStar Clinical Research Center, Washington D.C., District of Columbia
  - Medical Research Unlimited, Aventura, Florida
  - Internal Medicine Associates, Fort Myers, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Children's Clinic, Tallahassee, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - St. James Diabetes Center, Chicago Heights, Illinois
  - Indiana University Outpatient Clinical Research, Indianapolis, Indiana
  - University of Maryland Joslin Diabetes Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Grand Rapids Associated Interns, Grand Rapids, Michigan
  - Radiant Research, St Louis, Missouri
  - Mercury Street Medical, Butte, Montana
  - UNC Diabetes Care Center, Durham, North Carolina
  - Ohio State Univ.-Division of Endocrinology, Diabetes, Columbus, Ohio
  - Radiant Research, Portland, Oregon
  - Physicians for Clinical Research, Camp Hill, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - North Texas Clinical Research, Irving, Texas
  - Private Practice, Lufkin, Texas
  - Rainier Clinical Research Center, Renton, Washington

REFERENCES:
- [Derived] Herrmann K, Frias JP, Edelman SV, Lutz K, Shan K, Chen S, Maggs D, Kolterman OG. Pramlintide improved measures of glycemic control and body weight in patients with type 1 diabetes mellitus undergoing continuous subcutaneous insulin infusion therapy. Postgrad Med. 2013 May;125(3):136-44. doi: 10.3810/pgm.2013.05.2635. PMID 23748514